CLINICAL TRIAL: NCT06173609
Title: Long Left Internal Mammary Artery Patch on Left Anterior Descending Coronary Artery in Coronary Artery Bypass Grafting
Brief Title: Long LIMA Patch on Left Anterior Descending Coronary Artery in CABG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwan Ahmed Mohamed, Doctor, Assiut University
Other Study IDs: Long LIMA patch in CABG
Record Dates: First submitted 2023-12-08; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: CAD; LIMA; CABG
Keywords: CABG; LIMA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: CABG — During coronary artery bypass surgery, the surgeon removes a piece of blood vessel from the leg, chest, arm, or belly. Then, the surgeon uses that piece of blood vessel (called a "graft") to reroute blood around the blocked artery.

SUMMARY:
To assess the effect of LIMA patch as a method for the reconstruction on diffusely diseased LAD in the early and midterm outcomes

DETAILED DESCRIPTION:
It is well-known that coronary artery bypass graft (CABG) surgery significantly increases life expectancy, so complete myocardial revascularization should be the main goal of the surgical intervention process (1). During coronary artery bypass surgery, the surgeon removes a piece of blood vessel from the leg, chest, arm, or belly. Then, the surgeon uses that piece of blood vessel (called a "graft") to reroute blood around the blocked artery. The surgery is called "bypass surgery" because it bypasses the blockage Complete revascularization in CABG is crucial to improve early and late outcomes after surgery. Conventional procedures cannot achieve satisfactory results in severely diseased left anterior descending coronary artery .

Endarterectomy for severely atherosclerotic coronary artery disease (CAD) has a higher surgical risk and poor late outcomes . Reconstruction of diffusely diseased LAD with left internal mammary artery (LIMA) on-lay patch has less risk and complications than endarterectomy technique Ogus and colleagues used LIMA on-lay patches for the reconstruction of LAD based on the superior patency rate of the LIMA over other techniques which are more time-consuming. According to Lüscher and colleagues , the advantage of LIMA on-lay patch is to provide better vasomotor function and adjust the flow rate in proportion to the distal runoff.

In the recent study by Rezk etal., reported that , LAD reconstruction with a LIMA patch could have a better short-term outcome than other techniques as saphenous vein patch without an endarterectomy for a diffusely diseased left anterior descending coronary artery.

ELIGIBILITY:
Inclusion Criteria:

* Any patient male,( or female) and his(or her) age from 30-90 years have Ischemic Heart Disease for CABG with diffusely diseased LAD.

Exclusion Criteria:

* Any patient performed open heart surgery before

Ages: 30 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Perioperative data values were coded, processed and collected in tables. Qualitative data were described using number and percent. Quantitative data were described using median and standard deviation. Statistical significance was assumed if a p value of 0.05 or less was achieved.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
assess the effect of LIMA patch as a method for the reconstruction on diffusely diseased LAD in the early and midterm outcomes | first week postoperative
  asses postoperative new arrhythmia//use of Inotropes// second session of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Abdelrahman, professor, Study Chair — Professor of Cardiothoracic surgery; Ahmed Mohamed Taha, professor, Principal Investigator — Professor of Cardiothoracic surgery; Mohammed Hasan Osman, professor, Study Director — Professor of General surgery Maxillofacial surgery

REFERENCES:
- [Background] Todorov IP, Todorova ZP, Nikolov DP. Angioplasty balloon occlusion of LIMA graft in reoperations of patients with prosthetic valve endocarditis and patent LIMA-LAD graft. Kardiochir Torakochirurgia Pol. 2022 Dec;19(4):199-204. doi: 10.5114/kitp.2022.122089. Epub 2022 Dec 24. PMID 36643344
- [Background] Yang T, Yuan X, Li B, Zhao S, Sun H, Lu M. Long-term outcomes after coronary artery bypass graft with or without surgical ventricular reconstruction in patients with severe left ventricular dysfunction. J Thorac Dis. 2023 Apr 28;15(4):1627-1639. doi: 10.21037/jtd-22-1214. Epub 2023 Mar 23. PMID 37197557